CLINICAL TRIAL: NCT03351816
Title: Impact of New Biomarkers on the Maintenance of Sinus Rhythm After Cardioversion or Ablation of Atrial Fibrillation
Brief Title: Impact of New Biomarkers on Maintenance of Sinus Rhythm After Cardioversion or Ablation of Atrial Fibrillation
Acronym: Biorhythm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-A00731-52
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electric Countershock

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardioversion group (Experimental): Patients with persistent atrial fibrillation who are oriented for cardioversion in the course of routine care.
  Interventions: Procedure: Cardioversion
- Ablation group (Experimental): Patients with persistent or paroxystic atrial fibrillation who are oriented for ablation of AF in the course of routine care.
  Interventions: Procedure: Ablation of atrial fibrillation

INTERVENTIONS:
Procedure: Ablation of atrial fibrillation — Pulmonary vein isolation by radiofrequency or cryoablation.
  Arms: Ablation group
Procedure: Cardioversion — External electric shock delivery under general anesthesia.
  Arms: Cardioversion group

SUMMARY:
The Biorhythm study aims to investigate the utility of new biomarkers (e.g. MR proANP, ST2) measured pre-procedure for the prediction of procedural success in patients with atrial fibrillation undergoing cardioversion or ablation.

DETAILED DESCRIPTION:
This is a prospective, observational, multicentre study of patients with paroxystic or persistent atrial fibrillation scheduled to undergo cardioversion or ablation of AF in routine practice. Serum levels of MR proANP and ST2 pre-procedure will be measured to attempt to identify a threshold that carries prognostic value for procedural success (maintenance of sinus rhythm at one year).

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxystic or persistent atrial fibrillation for whom a decision to perform ablation is made.
* Patients with persistent atrial fibrillation for whom a decision to perform cardioversion is made.
* Patients with social security coverage, or beneficiary thereof.
* Patients who provide written informed consent.

Exclusion Criteria:

* Age <18 years or >80 years
* Patients with significant valvular heart disease defined as symptomatic aortic valve disease, severe aortic or mitral stenosis or tricuspid or mitral insufficiency grade 3/4 or 4/4
* Patients with pulmonary arterial hypertension >45 mmHg on echocardiography
* Patients with chronic respiratory disease, chronic obstructive pulmonary disease stage II, III or IV.
* Patients with a left ventricular ejection fraction <45%
* Patients with recent (<1 month) acute decompensation of heart failure
* Patients with recent (<1 month) acute coronary syndrome
* Anemia (hemoglobin <10 g/dL)
* Pregnant or lactating women
* Patients with anticipated poor compliance, as assessed by the study investigator
* Patients within the exclusion period of another clinical study
* Patients under legal guardianship

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Recurrent atrial fibrillation | 12 months
  Documented by ECG, Holter, telemetry, and lasting 30 seconds or more.
Recurrent atrial tachycardia | 12 months
  Documented by ECG, Holter, telemetry, and lasting 30 seconds or more.
Recurrent flutter | 12 months
  Documented by ECG, Holter, telemetry, and lasting 30 seconds or more.

SECONDARY OUTCOMES:
Recurrent atrial fibrillation | 3 months
  Documented by ECG, Holter, telemetry, and lasting 30 seconds or more.
Recurrent atrial tachycardia | 3 months
  Documented by ECG, Holter, telemetry, and lasting 30 seconds or more.
Recurrent flutter | 3 months
  Documented by ECG, Holter, telemetry, and lasting 30 seconds or more.
Palpitations | 12 months
  Any episode of palpitation occurring during follow-up
Hospitalization | 12 months
  Hospital admission related to atrial fibrillation, atrial tachycardia or flutter during follow-up
Repeat ablation | 12 months
  Need for repeat ablation during follow-up in patients who underwent ablation of AF
Cardioversion | 12 months
  Need for electric or medical cardioversion during follow-up (all patients, regardless of initial intervention type)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Meneveau, MD, PhD, Study Director — Centre Hospitalier Universitaire de Besancon
Locations (3):
- France (3):
  - University Hospital Jean Minjoz, Besançon
  - CHU François Mitterand, Dijon
  - CHU Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Badoz M, Serzian G, Favoulet B, Sellal JM, De Chillou C, Laurent G, Ecarnot F, Bardonnet K, Seronde MF, Schiele F, Meneveau N. MR-proANP, sST2, BNP and sinus rhythm maintenance 1 year after electrical cardioversion for atrial fibrillation. BMC Cardiovasc Disord. 2025 Aug 29;25(1):640. doi: 10.1186/s12872-025-05052-5. PMID 40883706
- [Derived] Badoz M, Serzian G, Favoulet B, Sellal JM, De Chillou C, Hammache N, Laurent G, Mebazaa A, Ecarnot F, Bardonnet K, Seronde MF, Schiele F, Meneveau N. Impact of Midregional N-Terminal Pro-Atrial Natriuretic Peptide and Soluble Suppression of Tumorigenicity 2 Levels on Heart Rhythm in Patients Treated With Catheter Ablation for Atrial Fibrillation: The Biorhythm Study. J Am Heart Assoc. 2021 Jul 6;10(13):e020917. doi: 10.1161/JAHA.121.020917. Epub 2021 Jun 30. PMID 34187182